CLINICAL TRIAL: NCT06585787
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Safety and Efficacy of KarXT for the Treatment of Psychosis Associated With Alzheimer's Disease
Brief Title: A Study to Evaluate KarXT as a Treatment for Psychosis Associated With Alzheimer's Disease (ADEPT-4)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN012-0056
Record Dates: First submitted 2024-08-30; First posted 2024-09-19 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; AD; ADEPT4; ADEPT-4; KarXT; Psychosis
MeSH Terms: conditions — Alzheimer Disease; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: KarXT
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510
  Arms: KarXT
Drug: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of KarXT in adult participants with mild to severe Alzheimer's Disease (AD) with moderate to severe psychosis related to AD.

ELIGIBILITY:
Inclusion Criteria

* Patients who are 55 to 90 years of age, inclusive, at the time of Screening (Visit 1).
* Patients who are diagnosed with AD based on the 2024 National Institute on Aging - Alzheimer's Association criteria with AD biomarker confirmation.
* Patient must have a magnetic resonance imaging (MRI) or computed tomography (CT) scan of the brain (completed within the past 5 years) taken during or subsequent to the onset of dementia to rule out other central nervous system (CNS) disease that could account for the dementia syndrome, eg, major stroke, neoplasm, subdural hematoma.
* Patient must have a history of psychotic symptoms (meeting International Psychogeriatric Association criteria) for at least 2 months prior to Screening (Visit 1) (participants may or may not have symptoms of agitation).

Exclusion Criteria

- Patients will not be able to participate if they have:.

i) Psychotic symptoms that are primarily attributable to a condition other than the AD causing the dementia, eg, schizophrenia, schizoaffective disorder, delusional disorder, or mood disorder with psychotic features.

ii) History of major depressive episode with psychotic features during the 12 months prior to Screening, or history of bipolar disorder, schizophrenia, or schizoaffective disorder.

iii) Patients are not able to participate if they have certain safety concerns, including certain laboratory test irregularities.

* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2026-09-21 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Neuropsychiatric Inventory-Clinician: Hallucinations and Delusions (NPI-C: H+D) score | Up to Week 14

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impressions-Severity (CGI-S) scale | Up to Week 14
Change from baseline in Neuropsychiatric Inventory-Clinician (NPI-C) Core score: Hallucination Domain | Up to Week 14
Change from baseline in NPI-C Core score: Delusion Domain | Up to Week 14
Change from baseline in NPI-C Core score: Agitation Domain | Up to Week 14
Change from baseline in NPI-C Core score: Aggression Domain | Up to Week 14
Change from baseline in NPI-C Agitation score | Up to Week 14
Change from baseline in NPI-C Core score: Caregiver Distress Scale | Up to Week 14
Number of participants with a ≥ 40% improvement from Baseline in NPI-C: H+D score | Up to Week 14
Change from baseline in Cohen- Mansfield Agitation Inventory-International Psychogeriatric Association (CMAI-IPA) total score | Up to Week 14
Change from baseline in Cohen- Mansfield Agitation Inventory (CMAI) total score | Up to Week 14
Number of participants with Adverse Events (AEs) | Up to Week 14
Number of participants with Treatment-Emergent Adverse Events (TEAEs) | Up to Week 14
Number of participants with Serious Adverse Events (SAEs) | Up to Week 14
Number of participants with TEAEs leading to study withdrawal | Up to Week 14
Number of participants with procholinergic symptoms | Up to Week 14
Number of participants with anticholinergic symptoms | Up to Week 14
Number of participants with AEs of Special Interest (AESIs) | Up to Week 14
Barnes Akathisia Rating Scale (BARS) Score | Up to Week 14
Abnormal Involuntary Movement Scale (AIMS) Score | Up to Week 14
Body Weight | Up to Week 14
Body Mass Index (BMI) | Up to Week 14
Number of participants with vital sign abnormalities | Up to Week 14
Number of participants with clinical laboratory abnormalities | Up to Week 14
Number of participants with 12-lead electrocardiogram (ECG) abnormalities | Up to Week 14
Number of participants with suicidal ideation as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS) | Up to Week 14
Cognition as assessed by the Mini-Mental State Examination (MMSE) | Up to Week 14
Cognition as assessed by the Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog-13) | Up to Week 14

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (272):
- United States (88):
  - Chandler Clinical Trials, LLC, Chandler, Arizona
  - Gilbert Neurology Partners - PLLC - Avacare, Gilbert, Arizona
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Scottsdale Clinical Trials, Scottsdale, Arizona
  - Advanced Research Center, Inc., Anaheim, California
  - Inland Psychiatric Medical Group (IPMG)-Chino, Chino, California
  - Long Beach Research Institute, LLC, Long Beach, California
  - USC - The Memory and Aging Center (MAC) - Alzheimer Disease Research Center (ADRC), Los Angeles, California
  - Local Institution - 1219, Los Angeles, California
  - ATP Clinical Research-302 W La Veta Ave, Orange, California
  - NRC Research Institute - Orange - PPDS, Orange, California
  - SC3 Research - Pasadena - 960 E. Green St, Pasadena, California
  - Prospective Research Innovations 8577 Haven Ave, Rancho Cucamonga, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Genesis Trust Research Group, Atlantis, Florida
  - Envision Trials LLC, Bonita Springs, Florida
  - JY Research Institute Inc, Cutler Bay, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Quantum Laboratories, Inc - West Palm Beach Office, Deerfield Beach, Florida
  - Integrity Clinical Research, LLC - 8000 NW 21st St, Doral, Florida
  - New Life Medical Research Center -3750 W 16th Ave, Hialeah, Florida
  - Research in Miami, Inc, Hialeah, Florida
  - Nexus Clinical Research Center- NRC, Homestead, Florida
  - K2 Medical Research - Lady Lake, Lady Lake, Florida
  - Homestead Associates in Research Inc, Miami, Florida
  - Premier Clinical Research Institute, Miami, Florida
  - Wellness Research Center Inc - Miami, Miami, Florida
  - A & D Doctor Center, Miami, Florida
  - Floridian Neuroscience Institute-1901 SW 1 St, Miami, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - MedOne Clinical Research LLC, Miami, Florida
  - My Community Research Center, Inc - 7480 Bird Rd, Miami, Florida
  - Future Care Solution LLC, Miami, Florida
  - Reliant Medical Research, Miami, Florida
  - Novel Clinical Research Center, LLC., Miami, Florida
  - Dade Research Center - Miami FL - 7600 SW 87th Ave, Miami, Florida
  - US Associates in Research Inc, Miami, Florida
  - Serenity Research Center, Miami, Florida
  - IMIC LLC- 9380 SW 150th Str, Miami, Florida
  - New Gen Health, Miami, Florida
  - Floridian Research Institute-1021 Ives Dairy Rd, Miami, Florida
  - High Quality Research, Miami, Florida
  - New Med Research, Miami Gardens, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Angels Clinical Research Institute - Miami Lakes - Palm Springs - PPDS, Miami Lakes, Florida
  - Aqualane Clinical Research, Naples, Florida
  - Sensible HealthCare, LLC, Ocoee, Florida
  - Nova Psychiatry, Orlando, Florida
  - Combined Research Orlando Phase I-IV LLC, Orlando, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Progressive Medical Research (Duplicate), Port Orange, Florida
  - Cordova Research Institute- Sweetwater, Sweetwater, Florida
  - Angels Clinical Research Institute Tampa - Palm Springs - PPDS, Tampa, Florida
  - Guardian Angel Research, Tampa, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Local Institution - 1233, Wellington, Florida
  - Premiere Research Institute at Palm Beach Neurology, PA, West Palm Beach, Florida
  - Agile Clinical Research Trials, LLC, Atlanta, Georgia
  - McLean Hospital, Belmont, Massachusetts
  - Tufts Medical Center - 800 Washington St - PPDS, Boston, Massachusetts
  - Boston Neuro Research Center, North Dartmouth, Massachusetts
  - Local Institution - 1250, South Dartmouth, Massachusetts
  - Elixia Health - Springfield - Elixia - PPDS, Springfield, Massachusetts
  - Neurobehavioral Medicine Group (NBMG), Bloomfield Township, Michigan
  - Precise Research Centers, Flowood, Mississippi
  - Advanced Memory Research Institute - CenExel - PPDS, Toms River, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - Local Institution - 1251, New Windsor, New York
  - Local Institution - 1231, Syracuse, New York
  - Local Institution - 1240, Syracuse, New York
  - Five Towns Neurology, PC, Woodmere, New York
  - Triad Clinical Trials - 515 College Rd, Greensboro, North Carolina
  - AMC Research, LLC - Flourish - PPDS, Matthews, North Carolina
  - Local Institution - 5005, Morehead City, North Carolina
  - West Clinical Research, Morehead City, North Carolina
  - Local Institution - 1252, Shelby, North Carolina
  - Ohio State University, Columbus, Ohio
  - Insight Clinical Trials LLC - Independence, Independence, Ohio
  - The Rivus Wellness & Research Institute, Oklahoma City, Oklahoma
  - Alzheimer's Disease and Memory Disorders Center at Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt Psychiatric Hospital, Nashville, Tennessee
  - Epic Medical Research LLC - DeSoto - HyperCore - PPDS, DeSoto, Texas
  - Advanced Neuro Research Center - El Paso, El Paso, Texas
  - AIM Trials, Plano, Texas
  - Glenn Biggs Institute for Alzheimer's & Neurodegenerative Diseases, San Antonio, Texas
  - R & H Clinical Research-3727 Greenbriar Dr, Stafford, Texas
  - Conquest Research - Arlington, Arlington, Virginia
  - Local Institution - 1253, Bellevue, Washington
- Argentina (9):
  - CINME S.A. - Centro de Investigaciones Metabólicas - Viamonte 2213/2215, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5005, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5001, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Local Institution - 5008, Rosario, Santa Fe Province
  - Local Institution - 5002, Buenos Aires
  - Local Institution - 5009, Buenos Aires
  - Local Institution - 5006, Buenos Aires
  - Local Institution - 5003, Córdoba
  - Local Institution - 5007, San Rafael
- Belgium (5):
  - UZ Brussel - PPDS, Jette, Brussels Capital
  - AZ Delta- Campus Rumbeke, Roeselare, West-Vlaanderen
  - ANIMA Research Center - PPDS, Alken
  - Local Institution - 2807, Bruges
  - AZ Groeninge, Kortrijk
- Brazil (7):
  - L2 Ip - Instituto de Pesquisas Clinicas Ltda - ME, Brasília, Federal District
  - CPQuali Pesquisa Clínica Sao Paulo, São Paulo, São Paulo
  - BR Trials - Pesquisa Clínica, São Paulo, São Paulo
  - Local Institution - 6207, São Paulo, São Paulo
  - Clinilive, São Paulo, São Paulo
  - Ruschel Medicina, Rio de Janeiro
  - Instituto de Psiquiatria HC FMUSP, São Paulo
- Bulgaria (4):
  - Medical Center Intermedica OOD, Sofia, Sofia-Grad
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD-66 Peshtersko Shosse blvd, Plovdiv
  - University Multiprofile Hospital For Active Treatment Kanev AD, Rousse
  - Medical Center Medika 2005 - Branch Sofia, Sofia
- China (20):
  - Local Institution - 7004, Beijing, Beijing Municipality
  - Local Institution - 7005, Beijing, Beijing Municipality
  - Local Institution - 7025, Beijing, Beijing Municipality
  - Local Institution - 7015, Chongqing, Chongqing Municipality
  - Local Institution - 7008, Guangzhou, Guangdong
  - Local Institution - 7016, Guangzhou, Guangdong
  - Local Institution - 7003, Shenzhen, Guangdong
  - Local Institution - 7013, Nanjing, Jiangsu
  - Local Institution - 7024, Nanjing, Jiangsu
  - Local Institution - 7023, Zhenjiang, Jiangsu
  - Local Institution - 7001, Shanghai, Shanghai Municipality
  - Local Institution - 7028, Shanghai, Shanghai Municipality
  - Local Institution - 7026, Shanghai, Shanghai Municipality
  - Local Institution - 7002, Chengdu, Sichuan
  - Local Institution - 7019, Tianjin, Tianjin Municipality
  - Local Institution - 7020, Hangzhou, Zhejiang
  - Local Institution - 7021, Hangzhou, Zhejiang
  - Local Institution - 7006, Hangzhou, Zhejiang
  - Local Institution - 7027, Changsha
  - Local Institution - 7022, Kunming
- Croatia (5):
  - Local Institution - 4106, Zagreb, City of Zagreb
  - Polyclinic Neuron, Zagreb, City of Zagreb
  - University Hospital Center Zagreb, Zagreb, City of Zagreb
  - Klinika za psihijatriju Vrapce, Zagreb, City of Zagreb
  - Psychiatric Clinic Sveti Ivan, Zagreb, City of Zagreb
- France (4):
  - Institut Claude Pompidou, Nice, Alpes-Maritimes
  - CHRU de Tours - Hôpital Bretonneau, Tours, Indre-et-Loire
  - Local Institution - 2512, Toulouse
  - CHU de Toulouse- Gerontopole, Toulouse
- Germany (5):
  - Local Institution - 2407, Böblingen, Baden-Wurttemberg
  - Universitatsklinikum des Saarlandes, Homburg, Saarland
  - Local Institution - 2406, Berlin
  - NeuroCentrum Odenwald, Erbach im Odenwald
  - Universitätsklinikum Frankfurt, Frankfurt am Main
- Greece (5):
  - Henry Dunant Hospital Center, Athens, Attica
  - University General Hospital ''ATTIKON'' - General Hospital of West Attica H AGIA VARVARA, Chaidari, Athens, Attica
  - General Oncology Hospital of Kifissia ''Agioi Anargyroi'', Kalyftaki-N. Kifissia, Attica
  - PAGNI-University General Hospital of Heraklion, Heraklion, Irakleio
  - 424 General Military Training Hospital-Outpatient Psychiatric Department, Thessaloniki
- Hungary (5):
  - Psychotech Kft., Pécs, Baranya
  - Local Institution - 4610, Szeged, Csongrád megye
  - Clinexpert Gyöngyös Kft., Gyöngyös, Heves County
  - Semmelweis Egyetem Pszichiátriai és Pszichoterápiás Klinika, Budapest
  - Eszak-budai Szent Janos Centrumkorhaz, Budapest
- India (6):
  - Local Institution - 7401, Nagpur, Maharashtra
  - Local Institution - 7405, Chandigarh, Punjab
  - Local Institution - 7406, Ajmer, Rajasthan
  - Local Institution - 7403, Hyderabad
  - Local Institution - 7404, Kolkata
  - Local Institution - 7402, Varanasi
- Israel (4):
  - Hadassah Medical Center- Ein Kerem - PPDS, Jerusalem, Jerusalem
  - The Barzilai University Medical Center, Ashkelon, Tel Aviv
  - Rabin Medical Center - PPDS, Petah Tikva
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan
- Italy (8):
  - Local Institution - 2325, Salerno, Campania
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I - Viale del Policlinico 155, Rome, Lazio
  - IRCCS San Raffaele- Via di Val Cannuta 250, Rome, Lazio
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Lombardy
  - Auxologico IRCCS - Auxologico San Luca, Milan, Lombardy
  - ASL Biella - Ospedale degli Infermi, Ponderano (Biella), Piedmont
  - Local Institution - 2321, Rome, Roma
  - Azienda Ospedaliero-Universitaria Sant'Andrea, Roma
- Japan (27):
  - Iizuka Memorial Hospital, Iizuka, Fukuoka
  - Southern TOHOKU Medical Clinic, Kōriyama, Fukushima
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-Shi, Hyōgo
  - Memory Clinic Toride, Toride-shi, Ibaraki
  - Kagawa Prefectural Central Hospital, Takamatsu, Kagawa-ken
  - Hatano Kousei Hospital, Hadano, Kanagawa
  - Koukan Clinic, Kawasaki-Shi, Kanagawa
  - Tsurumi Nishii Hospital, Yokohama, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - National Hospital Organization Utano National Hospital, Kyoto, Kyoto
  - National Hospital Organization Miechuo Medical Center, Tsu, Mie-ken
  - Asakayama General Hospital, Sakai, Osaka
  - Shin-Abuyama Hospital, Takatsuki, Osaka
  - Local Institution - 7510, Kanzaki-Gun Yoshinogari-Cho, Saga-ken
  - National Hospital Organization Saitama Hospital, Wako-Shi, Saitama
  - NHO Tokushima Medical Center West, Yoshinogawa, Tokushima
  - Tokyo Angel Hospital, Hachiōji, Tokyo
  - Sangenjaya Nakamura Mental Clinic, Setagaya-Ku, Tokyo
  - Kurumi Clinic, Setagaya-Ku, Tokyo
  - Tokyo Metropolitan Matsuzawa Hospital, Setagaya-Ku, Tokyo
  - Tokyo Metropolitan Geriatric Hospital, tabashi City, Tokyo
  - Local Institution - 7515, Fukuoka
  - Funairi nou clinic, Hiroshima
  - Yuge Neuropsychiatric Hospital, Kumamoto
  - Tsutsujimental Hospital, Tatebayashi
- Poland (8):
  - Centrum Medyczne HCP Szpital im. Jana Pawla II, Poznan, Greater Poland Voivodeship
  - Uniwersyteckie Centrum Kliniczne w Gdansku - Smoluchowskiego 17, Gdansk, Pomeranian Voivodeship
  - Osrodek Badan Klinicznych BD Research Sp. z o.o. - Andersa 3, Iława, Warmian-Masurian Voivodeship
  - Local Institution - 4213, Kielce
  - Pro Salus Sp. z o.o.sp. k, Lodz
  - NZOZ NEUROMED M. I M. Nastaj Spolka Partnerska -Lublin, Lublin
  - Local Institution - 4216, Sochaczew
  - 4 Wojskowy Szpital Kliniczny z Poliklinika SP ZOZ, Wroclaw
- Portugal (6):
  - ULS do Alto Ave, EPE - Hospital da Senhora da Oliveira Guimarães, Guimarães, Braga District
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon, Lisbon District
  - Campus Neurológico Sénior, Torres Vedras, Lisbon District
  - ULS de Matosinhos, EPE - Hospital Pedro Hispano, Matosinhos Municipality, Porto District
  - ULS de Santa Maria,EPE - Hospital de Santa Maria - PPDS, Lisbon
  - Local Institution - 2706, Lisbon
- Puerto Rico (5):
  - Santa Cruz Behavioral PSC, Bayamón
  - CDT Grupo Medico San Pablo Inc., Bayamón
  - Instituto De Neurologia Dra. Ivonne Fraga,Psc, San Juan
  - Barbara Diaz Hernandez MD Research Inc, San Juan
  - Local Institution - 1305, San Juan
- Romania (6):
  - CMI Dr. Buhas Ramocea Elena Daniela - Cabinet Medical de Psihiarie, Oradea, Bihor County
  - Prof Dr Alexandru Obregia Clinical Psychiatric Hospital- Centrul de Sanatate Mintala, Bucharest
  - Cai Ferate Clinical Hospital Constanta, Constanța
  - Institutul Privat de Cercetări Melchisedec pentru Boli Autoimune, Ereditare și Rare -I.P.C.M, Craiova
  - Local Institution - 4905, Iași
  - S.C. Carpe Diem SRL, Sibiu
- Serbia (7):
  - University Clinical Center of Serbia - Dr Subotica 6 - PPDS, Belgrade, Belgrade
  - Clinical Hospital Center Dragisa Misovic Dedinje, Belgrade
  - Military Medical Academy, Belgrade
  - Special Hospital for Psychiatric Diseases "Gornja Toponica", Gornja Toponica
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
- Slovakia (6):
  - Univerzitna nemocnica L Pasteura Kosice-Rastislavova 43, Košice, Košice Region
  - MUDr. Beata Dupejova - Neurologicka Ambulancia s.r.o, Banská Bystrica
  - KONZILIUM s.r.o, Dubnica nad Váhom
  - EPAMED s.r.o, Košice
  - Psychiatrická nemocnica Philippa Pinela Pezinok, Pezinok
  - Crystal Comfort, s.r.o., Vranov nad Topľou
- South Korea (12):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggido
  - Yongin Severance Hospital, Yonsei University Health System, Yongin-si, Gyeonggido
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Seoul Hospital, Seoul, Seoul Teugbyeolsi
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul Teugbyeolsi
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Yeongdeungpo-gu, Seoul Teugbyeolsi
  - Hallym University Chuncheon Sacred Heart Hospital, Gangwon-do
  - Seoul National University Hospital, Seoul
  - Local Institution - 7219, Seoul
  - Local Institution - 7203, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (8):
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Local Institution - 2213, Málaga, Málaga
  - Hospital Universitari Santa Maria, Lleida
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario De Salamanca, Salamanca
  - Hospital Victoria Eugenia, Seville
  - Hospital Universitario Rio Hortega, Valladolid
  - Local Institution - 2206, Zaragoza
- Turkey (Türkiye) (6):
  - Ondokuz Mayis Universitesi Tip Fakultesi Hastanesi, Atakum, Samsun
  - Hacettepe University Medical Faculty, Ankara
  - Eskisehir Osmangazi Universitesi Tip Fakultesi Hastanesi, Eskişehir
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Arastirma ve Uygulama Hastanesi, Izmir
  - IEU Medical Point Izmir Hastanesi, Izmir
- Ukraine (6):
  - Local Institution - 8001, Vinnytsia, Vinnytsia Oblast
  - Local Institution - 8003, Khmelnytskyi
  - Local Institution - 8006, Lviv
  - Local Institution - 8004, Smila
  - Local Institution - 8005, Uzhhorod
  - Local Institution - 8002, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06585787.html